CLINICAL TRIAL: NCT06776211
Title: Effectiveness of Virtual Reality and Low-Reality Simulation Application in Neonatal Resuscitation Skills Training
Brief Title: Effectiveness of VR and LR Applications in Newborn Resuscitation Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Leyla Kaya, Assoc. Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17.12.2024-34256
Record Dates: First submitted 2024-12-26; First posted 2025-01-15 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Virtual Reality; Neonatal Resuscitation; Simulation
Keywords: Neonatal Resuscitation; midwifery students; virtual reality; Simulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Simulation (Experimental): Virtual reality simulation application:
  The video content to be used in the virtual reality-based application was created by researchers from the Ministry of Health of the Republic of Turkey, General Directorate of Public Health, Neonatal Resuscitation Programme (NRP) Practitioner Certified Training Programme. The duration of the video was planned not to exceed 10 minutes in order not to reduce the interest and attention span.
  Interventions: Behavioral: Virtual Reality Simulation
- Low-Reality Simulation (Experimental): Low reality simulation application: The low reality simulation application to be used will use a neonatal model as a teaching aid, with human anatomy and functional features designed to simulate neonatal resuscitation applications.
  Interventions: Behavioral: Low-Reality Simulation

INTERVENTIONS:
Behavioral: Virtual Reality Simulation — Virtual reality simulation application:
  The video content to be used in the virtual reality-based application was created by researchers from the Ministry of Health of the Republic of Turkey, General Directorate of Public Health, Neonatal Resuscitation Programme (NRP) Practitioner Certified Training Programme. The duration of the video was planned not to exceed 10 minutes in order not to reduce the interest and attention span.
  Arms: Virtual Reality Simulation
Behavioral: Low-Reality Simulation — Low reality simulation application: The low reality simulation application to be used will use a neonatal model as a teaching aid, with human anatomy and functional features designed to simulate neonatal resuscitation applications.
  Arms: Low-Reality Simulation

SUMMARY:
This research was designed to investigate the effectiveness of virtual reality and low reality simulation applications in neonatal resuscitation skills training.

DETAILED DESCRIPTION:
The research universe will consist of fourth year students studying at the Department of Midwifery, Hamidiye Faculty of Health Sciences (HSBF), Health Sciences University (SBU) in the academic year 2024-2025 (N: 80).

In the preparation phase of the research, the literature on neonatal resuscitation will be reviewed by the researchers and the topic will be translated into an 8-week power point presentation. The 2-hour training content will also include case discussion and video demonstration of skills.

Randomisation of the study Students who volunteer to participate in the study will be allocated to the intervention and control groups using computerised simple random sampling. The study will use computer-assisted randomisation and students will be randomly assigned to the intervention and control groups using the program with the URL address https://www.randomizer.org.

By dividing the students into two groups as Virtual Reality Simulation Application and Low Reality Simulation Application, the students will be given an "Introductory Information Form", "Neonatal Resuscitation Information Form" and "Neonatal Resuscitation Skill Assessment Form".

In this planned experimental pre-test and post-test design and control group study, students were divided into Virtual Reality (n₁=40) and Low Reality Simulation (n₂=40) groups.

Each stage of the study and any applications to be made will be explained and a voluntary informed consent form will be obtained from each student.

Students will be assessed 4 weeks after the pre-test, post-test and application.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the research.
* Be an active student in the 4th year of the Midwifery Department of Hamidiye Health Sciences Faculty, University of Health Sciences.
* Attend theoretical classes regularly.

Exclusion Criteria:

* Being a passive student in the 4th year of the Midwifery Department of Hamidiye Health Sciences Faculty, University of Health Sciences.
* Not meeting the inclusion criteria.
* Having attended the Neonatal Resuscitation Certificate Training or Course.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Famale
Enrollment: 80 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Neonatal Resuscitation Information Form | Pre-test, immediately after participants were assigned to groups
  This form, developed by researchers based on literature, includes questions designed to assess midwifery students' knowledge. The information form was also based on the General Directorate of Public Health's Neonatal Resuscitation Program (NRP) Certified Practitioner Training Program. The form consists of 30 questions and includes true/false responses. Percentage and frequency measurements will be used to evaluate the form. The final form was developed based on expert opinion.
Neonatal Resuscitation Information Form | immediately after the pre-test
  It is based on the General Directorate of Public Health, Newborn Resuscitation/Neonatal Resuscitation Programme (NRP) Certified Practitioner Training Programme.
Neonatal Resuscitation Information Form | Follow-up test, 4 weeks after the post-test was administered
  It is based on the General Directorate of Public Health, Newborn Resuscitation/Neonatal Resuscitation Programme (NRP) Certified Practitioner Training Programme.
Neonatal Resuscitation Skills Assessment Form | Pre-test, immediately after participants were assigned to groups
  It is based on the General Directorate of Public Health, Newborn Resuscitation/Neonatal Resuscitation Programme (NRP) Certified Practitioner Training Programme.
Neonatal Resuscitation Skills Assessment Form | immediately after the pre-test
  It is based on the General Directorate of Public Health, Newborn Resuscitation/Neonatal Resuscitation Programme (NRP) Certified Practitioner Training Programme.
Neonatal Resuscitation Skills Assessment Form | Follow-up test, 4 weeks after the post-test was administered
  It is based on the General Directorate of Public Health, Newborn Resuscitation/Neonatal Resuscitation Programme (NRP) Certified Practitioner Training Programme.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Kaya, PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No